CLINICAL TRIAL: NCT00065455
Title: Pilot Study on the Effect of Vitamin A Supplementation on Cone Function in Retinitis Pigmentosa
Brief Title: Investigating the Effect of Vitamin A Supplementation on Retinitis Pigmentosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030255; 03-EI-0255
Record Dates: First submitted 2003-07-23; First posted 2003-07-24 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-05-06

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis Pigmentosa; Vitamin A; ERG; RP
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Vitamin A

INTERVENTIONS:
Drug: Vitamin A

SUMMARY:
Retinitis pigmentosa (RP) is a collective term for a group of inherited retinal dystrophies that are a major cause of irreversible blindness. RP of some type occurs in approximately 1 out of 3500 persons in the United States(1). Gene mutations are responsible for the majority of RP. To date, mutations have been identified in 30 different genes linked to RP(2). The visual prognosis of RP is poor, since the gradual but relentless visual field loss leads eventually to some degree of blindness(3). Although no effective treatment for RP has been identified, participants supplemented with a daily oral dose of 15,000 IU vitamin A palmitate have shown, on average, a slower rate of deterioration of retinal function when the intervention is continued over several years(4). The purpose of this research is to determine whether administration of high oral doses of vitamin A can acutely improve cone photoreceptor function in RP participants as measured by electroretinography (ERG). In this interventional, non-randomized, prospective, pilot study, 5 participants will receive a daily oral dose of 50,000 IU of vitamin A palmitate for 4 weeks, followed by a maintenance dose of 15,000 IU daily for the subsequent 2 weeks. The primary efficacy outcome is a relative percentage change in ERG response amplitude subsequent to vitamin A supplementation. A secondary efficacy outcome is a relative percentage change in implicit time from pre- to post- vitamin A supplementation, with improvement specified as a shorter response implicit time. Other secondary outcomes will be improvements in visual field (Humphery, 10-2; sum of thresholds). Safety outcomes include visual fields, ETDRS visual acuity, intraocular pressure, serum vitamin A level and liver function tests.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is a collective term for a group of inherited retinal dystrophies that are a major cause of irreversible blindness. RP of some type occurs in approximately 1 out of 3500 persons in the United States. Gene mutations are responsible for the majority of RP. To date, mutations have been identified in 30 different genes linked to RP. The visual prognosis of RP is poor, since the gradual but relentless visual field loss leads eventually to some degree of blindness. Although no effective treatment for RP has been identified, participants supplemented with a daily oral dose of 15,000 IU vitamin A palmitate have shown, on average, a slower rate of deterioration of retinal function when the intervention is continued over several years. The purpose of this research is to determine whether administration of high oral doses of vitamin A can acutely improve cone photoreceptor function in RP participants as measured by electroretinography (ERG). In this interventional, non-randomized, prospective, pilot study, 10 participants (five with the RHO1 gene mutation and five without the mutation) will receive a daily oral dose of 50,000 IU of vitamin A palmitate for 4 weeks, followed by a maintenance dose of 15,000 IU daily for the subsequent 2 weeks. The primary efficacy outcome is a relative percentage change in ERG response amplitude subsequent to vitamin A supplementation. A secondary efficacy outcome is a relative percentage change in implicit time from pre- to post- vitamin A supplementation, with improvement specified as a shorter response implicit time. Other secondary outcomes will be improvements in visual field (Humphrey 10-2; sum of thresholds). Safety outcomes include visual fields, ETDRS visual acuity, intraocular pressure, serum vitamin A level and liver function tests.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants must meet the following criteria to participate in the study.

1. Men and women age 18 years of age and older. (Children will be excluded since there is a higher incidence of vitamin A toxicity in the pediatric population.)
2. Diagnoses of typical RP of all genetic subtypes (simplex, autosomal dominant, autosomal recessive, and X-linked), as determined primarily by abnormally reduced ERG rod response amplitudes that are relatively more affected than cone ERG amplitudes.
3. Mutation in the RHO1 gene as determined by genotyping.
4. Participants in whom flicker ERG can be measured reliably (standard flicker ERG amplitude greater than 2 microV).
5. Willingness to use contraception for the duration of the study.
6. Understood and signed consent.

EXCLUSION CRITERIA:

Participants with the following conditions will be excluded from study.

1. Participants with syndromic RP (i.e., Ushers syndrome).
2. Have abnormal liver function (greater than ULN ALT, AST, Alkaline Phosphate, or Total Bilirubin).
3. Hematocrit greater than 1.5 x ULN
4. Have abnormal kidney function (greater than1.5 mg/dL serum creatinine).
5. Currently or has taken greater than 15,000 IU/day vitamin A supplementation within 6 months of the first screening visit.
6. Is pregnant or lactating (due to evidence that sugests excessive intake of vitamin A could be tertogenic in humans and affect the content of breast milk).
7. Currently or has taken greater than 400 IU/day of vitamin E supplementation within 6 months of enrollment.
8. Vitamin A serum level exceeding 150 microg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11
Dates: Start 2003-07-17; Study Completion 2009-05-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Phelan JK, Bok D. A brief review of retinitis pigmentosa and the identified retinitis pigmentosa genes. Mol Vis. 2000 Jul 8;6:116-24. PMID 10889272
- [Background] Milam AH, Li ZY, Fariss RN. Histopathology of the human retina in retinitis pigmentosa. Prog Retin Eye Res. 1998 Apr;17(2):175-205. doi: 10.1016/s1350-9462(97)00012-8. PMID 9695792
- [Background] Huang PC, Gaitan AE, Hao Y, Petters RM, Wong F. Cellular interactions implicated in the mechanism of photoreceptor degeneration in transgenic mice expressing a mutant rhodopsin gene. Proc Natl Acad Sci U S A. 1993 Sep 15;90(18):8484-8. doi: 10.1073/pnas.90.18.8484. PMID 8378322